CLINICAL TRIAL: NCT00960037
Title: The Vitamin D Dose Response Curve in Obesity
Brief Title: Trial to Assess Response to Oral Vitamin D3 Supplementation in Obese Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Winthrop University Hospital (Other)
Responsible Party: Principal Investigator, John F. Aloia, MD, Director, Bone Mineral Research Center, Winthrop University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 08002
Record Dates: First submitted 2009-08-13; First posted 2009-08-17 (Estimated); Last update posted 2012-06-18 (Estimated); Status verified 2012-06

CONDITIONS: Obesity
Keywords: Vitamin D3; obesity; cholecalciferol
MeSH Terms: conditions — Obesity | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D (Experimental): Vitamin D3 supplementation based on baseline 25(OH)D level
  Interventions: Dietary Supplement: Oral vitamin D3
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo equivalent

INTERVENTIONS:
Dietary Supplement: Oral vitamin D3 — Vitamin D3 50-100 mcg capsule(depending on baseline serum 25(OH)D concentration) daily for 8 weeks.
  Arms: Vitamin D
Dietary Supplement: Placebo equivalent — One capsule daily for 8 weeks
  Arms: Placebo

SUMMARY:
This study is an extension of an earlier study of vitamin D supplementation conducted on normal weight individuals by Dr. John Aloia of the Bone Mineral Research Division at Winthrop University Hospital. The investigators plan to compare the response to vitamin D supplementation in obese individuals with the response already measured in normal weight individuals. The same dosing schedule of vitamin supplementation will be used as in the past. The doses used in the past have demonstrated safety in a number of trials, here at Winthrop as well as outside of Winthrop Hospital. Sixty study volunteers are planned for enrollment in the study. The study participants will mainly be recruited from a group of patients who have in the past been enrolled in the weight loss program at Winthrop Hospital. Each participant will be on vitamin D supplementation for a total of 8 weeks. Vitamin D blood levels will be measured before and at the end of the supplementation period. They will then be compared to see the change over time as a result of supplementation.

ELIGIBILITY:
Inclusion Criteria:

* obese adults aged 18-65 years and BMI>35

Exclusion Criteria:

* chronic medical illness (diabetes, malignancy, uncontrolled hypertension, kidney disease)
* subjects who have undergone bariatric surgery or currently enrolled in a medically supervised weight loss program
* BMI < 35
* pregnancy
* use of medication that influences vitamin D metabolism
* history of of hypercalcemia, hypercalciuria, nephrolithiasis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2009-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Change in serum 25(OH)D level from baseline. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John F Aloia, MD, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States